CLINICAL TRIAL: NCT07189338
Title: Apneic Oxygenation With High-flow Nasal Oxygenation After Preoxygenation With Noninvasive Ventilation Before Intubation in Hypoxemic Patients in Intensive Care Unit.
Acronym: APNEIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DR240020
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hypoxemic Acute Respiratory Failure
Keywords: IUC; Hypoxemic acute respiratory failure; HFNO
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Apneic oxygenation will be used with HFNO between the laryngoscopy and the successful intubation (study intervention).
  NIV alone will be used for the preoxygenation and hypoventilation phase until the laryngoscopy.
  Apneic oxygenation will be used with HFNO at the time of laryngoscopy after removing the facemask of NIV (with HFNO on and set with a flow at 60-70L.min-1, FiO2 1.0)
  Interventions: Procedure: Apneic oxygenation
- Control group (Other): The control group will receive usual care, i.e., no oxygen during the apneic phase (between the laryngoscopy and the success of the intubation procedure) During the preoxygenation and hypoventilation phase until laryngoscopy, NIV alone will be used as in the experimental group.
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Apneic oxygenation — * Preoxygenation will be performed using NIV for 3-5 min With nasal cannulas placed in standby beneath the patient's chin (with HFNO on and set with a flow at 60-70L.min-1, FiO2 1.0)
  * Rapide sequence induction
  * Hypoventilation phase will be continue for 1 min using NIV
  * At the time of laryngoscopy :
  After removing the facemask, the nasal cannulas of HFNO will be placed in the patient's nares then the laryngoscopy will be performed.
  * Use of capnography to confirm the success of procedure
  Arms: Experimental group
Procedure: Usual Care — * Preoxygenation will be performed using NIV for 3-5 min without HFNO
  * Rapide sequence induction
  * Hypoventilation phase will be continue using NIV for 1min
  * At the time of laryngoscopy :
  After removing the facemask, laryngoscopy will be performed without oxygen.
  * Use of capnography to confirm the success of procedure
  Arms: Control group

SUMMARY:
The aim of this clinical study is to assess whether apneic oxygenation with High-Flow Nasal Oxygen (HFNO) would decrease the incidence of severe hypoxemia compared to no apneic oxygenation during the intubation procedure (from the start of laryngoscopy to 5 minutes after successful intubation) in patients with hypoxemic acute respiratory failure.

The sponsor expects that apneic oxygenation (between the laryngoscopy and the success of intubation) with HFNO compared to no apneic oxygenation could decrease the risk of severe hypoxemia after intubation in hypoxemic critical ill patients.

Participants will be enrolled according to eligibility criteria and randomized into one of the following groups:

Experimental group : Apneic oxygenation will be used with HFNO between the laryngoscopy and the successful intubation (study intervention).

non-invasive ventilation (NIV) alone will be used for the preoxygenation and hypoventilation phase until the laryngoscopy. The nasal cannulas of HFNO will be placed on hold beneath the patient's chin (with HFNO on and set with a flow at 60-70L.min-1, FiO2 1.0) pending laryngoscopy began.

At the time of laryngoscopy: after removing the facemask of NIV, the nasal cannulas for HFNO will be placed in the patient's nares then the laryngoscopy will be performed.

Control group: The control group will receive usual care, i.e., no oxygen during the apneic phase (between the laryngoscopy and the success of the intubation procedure) During the preoxygenation and hypoventilation phase until laryngoscopy, NIV alone will be used as in the experimental group.

DETAILED DESCRIPTION:
Endotracheal intubation is often performed in intensive care unit (ICU). Severe complications (such as severe hypoxemia, hypotension, cardiac arrest) occur up to 50%. Severe hypoxemia is more frequent in patients with hypoxemia prior to intubation or during difficult intubation and could increase the risk of cardiac arrest.

The procedure of intubation includes, in order 1) a preoxygenation phase ending with iv administration of anesthetic drugs 2) a hypoventilation phase 3) an apneic phase beginning with laryngoscopy and ending with successful intubation 4) mechanical ventilation. Optimization of this procedure is essential.

Non-invasive ventilation (NIV) is recommended for preoxygenation in hypoxemic patients and this technique can maintain ventilation during the hypoventilation phase.

Apneic oxygenation is defined as the administration of oxygen during the apneic phase. The objective is to increase the duration of apnea without desaturation. In physiological studies and in the operating room, when apneic oxygen is used with standard oxygen (up to 15L/min) or high-flow nasal oxygenation (HFNO) (up to 70L/min and FiO2 at 1.0), the apnea length without desaturation can reach several minutes.

Several meta-analyses (with high heterogeneity between studies) found that apneic oxygenation (including standard oxygen or HFNO) in emergency intubation could decrease the risk of hypoxemia. In most studies that investigated the effect of HFNO as apneic oxygenation, HFNO was also used as a preoxygenation method. Thus, the different methods of preoxygenation could affect the real effect of apneic oxygenation.

Only one single-center study evaluated apneic oxygenation with HFNO after preoxygenation by NIV. In this study the lowest SpO2 during intubation procedure was significantly higher in the apneic oxygenation group. However, in this study the mask used for NIV was applied over the nasal cannulas of HFNO, which may have resulted in less efficient preoxygenation due to leakage.

Intubation rate for HFNO failure during acute respiratory failure is about 40% in ICU patients. The question of continuing HFNO or not during the apnea phase remains open. The experts suggest continuing HFNO during intubation (conditional recommendation, moderate certainty).

We hypothesized that apneic oxygenation (between the laryngoscopy and the success of intubation) with HFNO compared to no apneic oxygenation could decrease the risk of severe hypoxemia after intubation in hypoxemic critical ill patients.

In both groups, NIV will be used during the preoxygenation and hypoventilation phases.

Procedure of intubation will be standardized according to guidelines

* Preoxygenation will be performed using NIV through a facemask in both group

  1. Experimental group: The nasal cannulas of HFNO will be placed on hold beneath the patient's chin (with HFNO on and set with a flow at 60-70L.min-1, FiO2 1.0) pending laryngoscopy began.
  2. Control group: no HFNO
* Rapide sequence induction (etomidate or ketamine + succinylcholine or rocuronium)
* Hypoventilation phase will be continue in both groupe for 1min using NIV through a facemask
* At the time of laryngoscopy :

  1. Experimental group: after removing the facemask of NIV, the nasal cannulas for HFNO will be placed in the patient's nares then the laryngoscopy will be performed.
  2. Control group: After removing the facemask, laryngoscopy will be performed without oxygen.
* recommandation of using a videolaryngoscope with a bougie or stylet
* Use of capnography to confirm the success of procedure
* initiate or increase vasopressors if needed
* Initiation of long-term sedation
* Initiation protective ventilation

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in the ICU
* Indication of orotracheal intubation for Hypoxemic acute respiratory failure defined by:

  * One sign of acute respiratory distress (respiratory rate >25/min, dyspnea or the use of accessory respiratory muscle)
  * AND a PaO2/FiO2 ≤ 200 mmHg (measured or calculated FiO2) within 6 hours before the decision of intubation. For the calculation of FiO2, the FiO2 will be estimated by: FiO2 = 0.21 + 0.03 x (flow of oxygen) (Coudroy, Thorax 2020)
* Informed consent from the patient or relatives. An emergency procedure will be possible when necessary.

Exclusion Criteria:

* < 18 years old

  * Need for emergent intubation (i.e. cardiac arrest)
  * Contraindication to non-invasive ventilation for preoxygenation
  * Known allergy or contraindication to one of the induction drugs
  * SpO2 device specific for the study not available
  * Patients without any healthcare insurance scheme or not benefiting from it through a third party,
  * Persons under law protection, namely minors, pregnant or breastfeeding women, persons deprived of their liberty by a judicial or administrative decision
  * Previous participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe hypoxemia | from the start of laryngoscopy to 5 minutes after successful intubation
  The incidence of severe hypoxemia defined as the occurrence of at least one episode of oxygen saturation measured by pulse oximetry (SpO2) < 80%

SECONDARY OUTCOMES:
Incidence of prolonged severe hypoxemia | from the start of laryngoscopy to 5 minutes after successful intubation
  The incidence of prolonged severe hypoxemia defined by an SpO2 < 80% for more than 24 seconds
The highest and lowest SpO2 values during the procedure | from the start of laryngoscopy to 5 minutes after successful intubation
  The highest and lowest SpO2 values during the procedure
The occurrence of each immediate severe complications | from the start of laryngoscopy to 5 minutes after successful intubation
  The occurrence of each immediate severe complications including cardiovascular instability (systolic arterial blood pressure <65 mmHg at least once, new or increase need of vasopressors or fluid bolus >15 mL/kg), cardiac arrest, new onset cardiac arrhythmia (atrial fibrillation, ventricular tachycardia, bradycardia <30beats per minute).
The occurrence of each other adverse events | from the start of laryngoscopy to 5 minutes after successful intubation; At Day 28
  The occurrence of each other adverse events: difficult intubation (defined as a procedure requiring more than 2 laryngoscopy attempts before success), operator-reported aspiration between induction and intubation, dental injury, esophageal intubation, pneumothorax visualized on the follow-up chest X-ray as part of the patient's routine care.
Duration of laryngoscopy | From the 1st attempt to the successful intubation
  The duration of laryngoscopy will be compared in both group
Number of laryngoscopies | from the 1st attempt to the successful intubation
  The number of laryngoscopies will be compared in both group
Day-28 mortality | at Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Tours, Tours, France